CLINICAL TRIAL: NCT03664297
Title: Phase 1 Study to Evaluate the Tolerance and Pharmacokinetics of SHR1459 in Patients With Recurrentreplased/Refractory Mature B Cell Neoplasms Tumor
Brief Title: Tolerance and Pharmacokinetics of SHR1459 in Patients With Recurrent Replased/Refractory Mature B Cell Neoplasmstumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR1459-I-101
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Mature B Cell Neoplasms
Keywords: replased/refractory mature B cell neoplasms; BTK inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR1459 (Experimental): Oral administration, once a day, 28 days for a cycle, until the disease progression or the intolerable toxicity occurs.
  Interventions: Drug: SHR1459

INTERVENTIONS:
Drug: SHR1459 — SHR1459 will be administered continually till disease progression or unacceptable toxicity.
  Other Names: No other intervention

SUMMARY:
SHR1459 is a selective small molecule BTK inhibitor developed by Jiangsu Hengrui medicine Limited, by inhibiting the phosphorylation of BTK and down regulation of BCR signal transduction pathway, And then selectively inhibit the proliferation and migration of B cell tumor.

DETAILED DESCRIPTION:
SHR1459 is a selective small molecule BTK inhibitor developed by Jiangsu Hengrui medicine Limited, by inhibiting the phosphorylation of BTK and down regulation of BCR signal transduction pathway, And then selectively inhibit the proliferation and migration of B cell tumor. The objective of this phase 1 study is to evaluate the safety and tolerance of SHR1459 in patients with replaced/refractory mature B cell neoplasms, in order to determine the maximum tolerated dose (MTD) and recommended dose for phase 2 clinical study (RP2D);

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status [PS] score must be 0 or 1;
* Life expectancy ≥ 12 weeks;
* Mature B cell eoplasmss with histological or cytological diagnosis, including diffuse large B cell lymphoma (DLBCL), follicular lymphoma (FL) , chronic lymphocytic leukemia/Small lymphocytic lymphoma (CLL/SLL), Mantle cell lymphoma (MCL), Marginal zone lymphoma (MZL) and waldenstrom macroglobulinemia (WM);
* The function of bone marrow is basically normal;
* Renal function is basically normal;
* Hepatic function is basically normal.

Exclusion Criteria:

* Had received treatment with the compound of the same mechanism (BTK inhibitor);
* With infiltration of lymphoma central nervous system;
* Received autologous stem cell transplantation within 60 days before signing the informed consent, received allogeneic stem cell transplantation in 90 days (after allogeneic stem cell transplantation, if graft-versus-host disease appeared, it must be ≤ level 1, and if there was no prohibited medication, the screening could be performed);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (AEs) [Safety and Tolerability]) | through study completion, an average of about 6 months
  The incidence and severity of treatment-emergent AEs will be collected and the safety and tolerability of SHR1459 will be assessed
Recommended phase 2 dose (RP2D) | 28 days since the date of first dose
  Recommended phase 2 dose (RP2D) and/or maximum tolerated dose (MTD) will be established according to the incidence of dose-limiting toxicities (DLTs) of escalated doses of SHR1459

SECONDARY OUTCOMES:
Objective response rate (ORR) | every 8 weeks through study completion, an average of about 6 months
  Assess the response rate of subjects to the treatment of SHR1459
Duration of Response (DoR) | every 8 weeks through study completion, an average of about 6 months
  Assess the duration of complete/partial response after the treatment of SHR1459
Progression-free survival (PFS) | every 8 weeks through study completion, an average of about 6 months
  Assess the survival condition of the subjects after the treatment of SHR1459
Time to Response (TTR) | every 8 weeks through study completion, an average of about 6 months
  Assess time to response of SHR 1459 after treatment
Time to peak (Tmax) | Day 1 and Day 2 of the single dose
  Pharmacokinetics profile of a single dose SHR1459 and its metabolite (plasma): Time to peak (Tmax) of plasma concentration
Maximum plasma concentration (Cmax) | Day 1 and Day 2 of the single dose
  Pharmacokinetics profile of a single dose SHR1459 and its metabolite (plasma): Maximum plasma concentration (Cmax)
Halflife (T1/2) | Day 1 and Day 2 of the single dose
  Pharmacokinetics profile of a single dose SHR1459 and its metabolite (plasma): Halflife (T1/2)
Clearance/ bioavailability (CL/F) | Day 1 and Day 2 of the single dose
  Pharmacokinetics profile of a single dose SHR1459 and its metabolite (plasma): Clearance/ bioavailability (CL/F)
apparent volume of distribution/bioavailability (Vd/F) | Day 1 and Day 2 of the single dose
  Pharmacokinetics profile of a single dose SHR1459 and its metabolite (plasma): apparent volume of distribution/bioavailability (Vd/F)
Area under curve (AUC) | Day 1 and Day 2 of the single dose
  Pharmacokinetics profile of a single dose SHR1459 and its metabolite (plasma): Area under curve (AUC)
Area under curve, steady state (AUCss) | Day 1 of cycle 1 to day 1 of cycle 4 (28 days/cycle)
  Pharmacokinetics profile of a single dose SHR1459 and its metabolite (plasma): Area under curve, steady state (AUCss)
Maximum plasma concentration, steady state (Cmax,ss) | Day 1 of cycle 1 to day 1 of cycle 4 (28 days/cycle)
  Pharmacokinetics profile of a single dose SHR1459 and its metabolite (plasma): Maximum plasma concentration, steady state (Cmax,ss)
Time to peak, steady state (Tmax,ss) | Day 1 of cycle 1 to day 1 of cycle 4 (28 days/cycle)
  Pharmacokinetics profile of a single dose SHR1459 and its metabolite (plasma): Time to peak, steady state (Tmax,ss)
Halflife (T1/2) | Day 1 of cycle 1 to day 1 of cycle 4 (28 days/cycle)
  Pharmacokinetics profile of a single dose SHR1459 and its metabolite (plasma): Halflife (T1/2)
Apparent volume of distribution, steady state/bioavailability (Vss/F) | Day 1 of cycle 1 to day 1 of cycle 4 (28 days/cycle)
  Pharmacokinetics profile of a single dose SHR1459 and its metabolite (plasma): Apparent volume of distribution, steady state/bioavailability (Vss/F)
Clearance/ bioavailability (CL/F) | Day 1 of cycle 1 to day 1 of cycle 4 (28 days/cycle)
  Pharmacokinetics profile of a single dose SHR1459 and its metabolite (plasma): Clearance/ bioavailability (CL/F)
Accumulation index (Rac) | Day 1 of cycle 1 to day 1 of cycle 4 (28 days/cycle)
  Pharmacokinetics profile of a single dose SHR1459 and its metabolite (plasma): Accumulation index (Rac)

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Principal Investigator — Blood Institute of the Chinese Academy of Medical Sciences
Locations (1):
- Blood disease hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No